CLINICAL TRIAL: NCT03333616
Title: A Phase II Study of Nivolumab Combined With Ipilimumab for Patients With Advanced Rare Genitourinary Tumors
Brief Title: Nivolumab Combined With Ipilimumab for Patients With Advanced Rare Genitourinary Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Bradley A. McGregor, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-423
Record Dates: First submitted 2017-10-30; First posted 2017-11-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Genitourinary Cancer; Adrenocortical Carcinoma; Non-urothelial Bladder; Non-urothelial Upper Tract; Penile Cancer; Non-adenocarcinoma Prostate Cancer; Refractory Germ-cell; High Grade Neuroendocrine Carcinoma/Small Cell Carcinoma
Keywords: Genitourinary Cancer
MeSH Terms: conditions — Urogenital Neoplasms; Adrenocortical Carcinoma; Penile Neoplasms; Carcinoma, Small Cell | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab+Ipilimumab (Experimental): * Nivolumab and Ipilimumab are administered intravenously every 3 weeks for a total of 4 maximum doses. After combination therapy, nivolumab will be administered as monotherapy every 4 weeks.
  * Doses are determined per protocol.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilimumab — is an immunotherapy medication that stimulates the immune system to fight cancer cells throughout the body.
  Other Names: Yervoy
Drug: Nivolumab — Nivolumab binds to and blocks the activation of PD-1. This results in the activation of T-cells and cell-mediated immune responses against tumor cells
  Other Names: Opdivo

SUMMARY:
This research study is studying a combination of drugs as a possible treatment for rare genitourinary malignancies among four cohorts, bladder or upper tract carcinoma with variant histology, adrenocortical carcinoma, other rare genitourinary carcinomas and any genitourinary carcinoma with neuroendocrine differentiation. Given preliminary results, the study is being tested in additional patients with bladder or upper tract carcinoma with variant histology at this time while the adrenocortical carcinoma, other rare genitourinary malignancies arms have closed to accrual

-The names of the study drugs involved in this study are:

* Nivolumab
* Ipilimumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the combination of drugs works in treating a specific disease. "Investigational" means that the drugs are being studied.

The FDA (the U.S. Food and Drug Administration) has not approved nivolumab in combination with ipilimumab for this specific disease but the combination is approved for use in melanoma patients.

In this research study, the investigators are...

* Investigating the response of the participant's cancer to treatment with nivolumab plus ipilimumab,
* Assessing the safety of treatment with nivolumab and ipilimumab and
* Evaluating response and resistance to treatment by looking at the participant's tumor tissue and blood for markers to predict response and resistance to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2 within 28 days prior to registration (Appendix A).
* Unresectable advanced or metastatic ACC, non-urothelial bladder/upper tract cancer, non-adenocarcinoma prostate cancer, penile cancer, treatment refractory germ-cell tumor or a high grade neuroendocrine carcinoma/small cell carcinoma of any genitourinary site. Pure is defined as >90% and those with a portion of urothelial carcinoma or prostate adenocarcinoma may be included at discretion of the principal investigator. With variant histology in the primary, if metastatic biopsy shows pure variant histology, patient is eligible.
* at this time only the bladder and neuroendocrine cohorts are open
* Availability of Formalin-fixed, Paraffin-embedded (FFPE) archival tumor specimens, when available, and willingness of the subject to undergo mandatory fresh tumor biopsy prior to treatment initiation unless determined medically unsafe or not feasible.

  * The archival specimen, when available, must contain adequate viable tumor tissue.
  * The specimen may consist of a tissue block (preferred and should contain the highest grade of tumor) or at least 20 unstained serial sections. Fine-needle aspiration, brushings, cell pellet from pleural effusion, bone marrow aspirate/biopsy are not acceptable.
  * A mandatory biopsy at the time of radiographic progression will be requested from patients who have an initial response to treatment and then subsequently progress as determined by RECIST version 1.1.
* Measurable disease as defined by RECIST 1.1 within 28 days prior to registration.
* Demonstrate adequate organ function. All screening labs to be obtained within 28 days prior to first study treatment.

  * Hematological

    * White blood cell (WBC) ≥ 2000 cells/µL
    * Absolute Neutrophil Count (ANC) ≥ 1000 cells/µL
    * Platelet count (plt) ≥ 75,000/ µL
    * Hemoglobin (Hgb) ≥ 9 g/dL
    * Absolute lymphocyte count ≥ 500 cells/µL
  * Renal

    * Serum creatinine OR
    * Calculated creatinine clearance1 ≤ 1.5 x ULN ≥ 40 mL/min
  * Hepatic and Other

    * Bilirubin ≤ 1.5 × upper limit of normal (ULN)
    * AST2 ≤ 2.5 × ULN
    * ALT2 ≤ 2.5 × ULN
    * Alkaline Phosphatase2 ≤ 2.5 × ULN
    * Albumin > 2.5 g/dL
  * Coagulation

    * International Normalized Ratio (INR) or Prothrombin Time (PT)
    * Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 × ULN (unless on prophylactic or therapeutic dosing with low molecular weight heparin or warfarin)
* Females of childbearing potential must have a negative urine or serum pregnancy test within 28 days prior to registration. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months
* Females of childbearing potential and males must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 120 days after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study

Exclusion Criteria:

* Prior use of systemic checkpoint inhibitors (including PD-1, PD-L1, and CTLA-4 targeting agents) for the management of ACC, non-urothelial bladder cancer/upper tract, non-adenocarcinoma prostate cancer, penile cancer or treatment refractory germ-cell tumor is excluded
* Treatment with systemic immunosuppressive medications including but not limited to: prednisone, dexamethasone, cyclosporine, azathioprine, methotrexate, thalidomide, anti-tumor necrosis factor (TNF) agents within 2 weeks of first study dose.

  * Subjects who have received acute, low-dose systemic immunosuppressant medications may be enrolled (such as steroids for acute nausea or cancer-related pain ≤ 10 mg prednisone) maybe enrolled sooner than 2 weeks of first study dose.
  * Subjects with adrenal insufficiency on physiologic replacement doses of steroids may be enrolled (≤ 10 mg prednisone).
  * The use of inhaled, topical, ocular or intra-articular corticosteroids and mineralocorticoids are allowed.
* Treatment with chemotherapy, hormone therapy, or other investigational therapy within 3 weeks of first study doses. Patients with non-adenocarcinoma of the prostate who may be on luteinizing hormone-releasing hormone agonist/antagonist therapy may continue use. For ACC patients, hormonal agents (e.g mitotane) are allowed for the purpose to control endocrine-related symptoms when needed.
* Radiotherapy within 14 days of first study treatment with the exception of a single fraction of radiation administered for palliation of symptoms.
* Known active metastases to the brain, spinal cord or leptomeninges. Patients who are treated with radiotherapy, radiosurgery, or surgery and clinically stable for at least 2 weeks of first study treatment are eligible. Repeat imaging is not required to document treatment response.
* Malignancies other than ACC, non-urothelial bladder/upper tract cancer, non-adenocarcinoma prostate cancer, penile cancer, treatment refractory germ-cell tumor or genitourinary high grade neuroendocrine carcinoma/small cell carcinoma within 5 years of first study treatment with the exception of those with negligible risk of metastases or death and/or treated with expected curative outcome (included but not limited to carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer for patients with malignancies other than non-adenocarcinoma of the prostate, ductal carcinoma in situ of the breast, non-muscle invasive urothelial carcinoma of the bladder for patients with malignancies other than non-urothelial bladder cancer).
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion protein.
* Known hypersensitivity to any component of the nivolumab or ipilimumab product.
* Any active or recent history (within 6 months of first study dose) of autoimmune disease or syndrome that requires systemic corticosteroids (>10 mg daily prednisone equivalent) or immunosuppressive medications including but not limited to: myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, Wegner's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Subjects with vitiligo, controlled type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement therapy are permitted to enroll.
* Any condition requiring treatment with corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medication within 14 days of the first dose of study drug. Inhaled, topical, ocular or intra-articular corticosteroids and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Uncontrolled adrenal insufficiency.
* History of idiopathic pulmonary fibrosis, organized pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening imaging CT of the chest. History of radiation pneumonitis in the radiation field is permitted.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome.
* Active or chronic hepatitis B infection (defined as having a positive hepatitis B surface antigen (HBsAg) test at screening). Subject with past or resolved hepatitis B infection (defined as having a negative HBsAg test and positive antibody to hepatitis B core antigen test) are eligible. Hepatitis B viral DNA must be obtained in Subjects with positive hepatitis B core antibody prior to first treatment start.
* Active hepatitis C infection. Subjects positive hepatitis C antibody test are eligible if PCR is negative for hepatitis C viral DNA.
* Receipt of therapeutic oral or IV antibiotics within 2 weeks of first study treatment. Subjects receiving routine antibiotic prophylaxis (for dental extractions/procedures) are eligible.
* Active infection requiring systemic treatment.
* Significant cardiovascular disease such New York Heart Association (NYHA) class III or greater, myocardial infarction within the previous 3 months, unstable arrhythmias, unstable angina, need for cardiac angioplasty or stenting, coronary artery by-pass graft surgery, symptomatic peripheral vascular disease. Subjects with known coronary artery disease treated with stenting or coronary artery by-pass graft, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must be on a stable regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist when appropriate.
* Prolongation of the QTcF interval defined as > 450 msec for males and > 470 msec for females.
* Inadequately controlled hypertension (defined as systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg). Anti-hypertensive therapy to achieve these parameters is allowed.
* History of cerebrovascular accident or transient ischemic attack within 3 months of first study dose.
* Significant vascular disease (such as aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 3 months of first study dose.
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation) within 4 weeks of first study dose.
* History of symptomatic deep vein thrombosis or pulmonary embolism within 4 weeks of first study dose.
* History of abdominal or tracheoesophageal fistula or GI perforation within 6 months of first study treatment.
* Clinical signs or symptoms of GI obstruction or requirement of routine parenteral nutrition or tube feedings.
* Evidence of abdominal free air not explained by paracentesis or recent surgical procedure.
* Serious, non-healing or dehiscing wound or active ulcer.
* Major surgical procedure within 4 weeks of first study treatment.
* Presence of any toxicities attributed to prior anti-cancer therapy that are not resolved to grade 2 (CTCAE version 4.0) or baseline that could impose risk for serious complications before administration of study drug,
* Prior allogenic stem cell or solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Imaging will occur every 6-12 weeks study entry up until disease progression (up to 24 months)
  Radiologic disease assessment performed at 12 weeks after initial treatment and then every 6 or 12 weeks. These radiologic disease assessments are evaluated per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 guidelines. This will be conducted by cohort ((1) ACC, (2) Non-urothelial bladder/upper tract cancer and (3) other rare GU tumors)

SECONDARY OUTCOMES:
Objective Response Rate for all rare GU tumor types | Imaging will occur every 6-12 weeks study entry up until disease progression (up to 24 months)
  Radiologic disease assessment performed at 12 weeks after initial treatment and then every 6 or 12 weeks. These radiologic disease assessments are evaluated per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 guidelines. A pooled analysis of all tumor cohorts will be done as a secondary analysis.
Duration of Response | Imaging will occur every 6-12 weeks study entry up until disease progression (up to 24 months)
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, or death due to any cause) estimated using the method of Kaplan-Meir for all patients and by tumor cohorts. (((1) ACC, (2) Non-urothelial bladder/upper tract cancer and (3) other rare GU tumors)
Immune related objective response rate | Imaging will occur every 6-12 weeks study entry up until disease progression (up to 24 months)
  Radiologic disease assessment performed at 12 weeks after initial treatment and then every 6 or 12 weeks. These radiologic disease assessments are evaluated per Immune-Related Response Criteria (irRC) and will be analyzed for all patients any by tumor cohort ((1) ACC, (2) Non-urothelial bladder/upper tract cancer and (3) other rare GU tumors)
Progression-Free Survival for the total cohort and by tumor cohort | From start of treatment until date of death from any cause (average 24 months)
  PFS is measured from the start of treatment until the documented progression by RESIST criteria or death from any cause. This will be summarized using the method of Kaplan-Meir for all patients and by tumor cohorts. ((1) ACC, (2) Non-urothelial bladder/upper tract cancer and (3) other rare GU tumors)
Overall Survival for all patients and by tumor cohort | From start of treatment until date of death from any cause. (Average 24 months)
  OS is measured from the start of treatment until date of death from any cause and will be analyzed in all patients and by tumor cohorts ((1) ACC, (2) Non-urothelial bladder/upper tract cancer and (3) other rare GU tumors)
Safety and tolerability according to Common Terminology Criteria for Adverse Events (CTCAE). | Throughout the course of the study, approximately 24 months after study entry.
  All adverse events recorded during the trial will be summarized for the safety population.The incidence of events that are new or worsening from the time of first dose of treatment will be summarized according to system organ class and/or preferred term, severity (based on CTCAE version 4), type of adverse event, and relation to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley A McGregor, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - University of California, San Diego Moores Cancer Center, La Jolla, California
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McGregor BA, Campbell MT, Xie W, Farah S, Bilen MA, Schmidt AL, Sonpavde GP, Kilbridge KL, Choudhury AD, Mortazavi A, Shah AY, Venkatesan AM, Bubley GJ, Siefker-Radtke AO, McKay RR, Choueiri TK. Results of a multicenter, phase 2 study of nivolumab and ipilimumab for patients with advanced rare genitourinary malignancies. Cancer. 2021 Mar 15;127(6):840-849. doi: 10.1002/cncr.33328. Epub 2020 Nov 20. PMID 33216356